CLINICAL TRIAL: NCT05667298
Title: A Phase I Study of Organ-Preserving Endoscopic Resection & Adjuvant RADIO-immuno-chemotherapy for Esophageal Cancer (OPERA-RADIO)
Brief Title: Organ-Preserving Endoscopic Resection & Adjuvant RADIO-immuno-chemotherapy for Esophageal Cancer
Acronym: OPERARADIO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other); CancerCare Manitoba (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Biniam Kidane, Principal Investigator, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001
Record Dates: First submitted 2022-10-06; First posted 2022-12-28 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — 26S proteasome non-ATPase regulatory subunit 13; Chemoradiotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: The primary/preferred adjuvant therapy will be immunoradiotherapy (ARM1); however, if this combination is felt to be too high-risk for specific patients, the next preferred therapy will be immunotherapy without radiation (ARM1B). Some patients have medical conditions, i.e., severe auto-immune disease that prohibits them from receiving immunotherapy. In such patients, adjuvant therapy will be provided in the form of concurrent chemoradiotherapy (ARM2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjuvant Immunoradiotherapy (ARM1) and Adjuvant Immunotherapy (ARM1B) (Experimental): The primary/preferred adjuvant therapy will be immunoradiotherapy (ARM1); however, if this combination is felt to be too high-risk for specific patients, the next preferred therapy will be immunotherapy without radiation (ARM1B).
  Interventions: Drug: Adjuvant Immunoradiotherapy (ARM1) and Adjuvant Immunotherapy (ARM1B)
- Adjuvant chemoradiotherapy (Experimental): Some patients have medical conditions, i.e., severe auto-immune disease that prohibits them from receiving immunotherapy. In such patients, adjuvant therapy will be provided in the form of concurrent chemoradiotherapy (ARM2).
  Interventions: Drug: Adjuvant chemoradiotherapy

INTERVENTIONS:
Drug: Adjuvant Immunoradiotherapy (ARM1) and Adjuvant Immunotherapy (ARM1B) — Durvalumab treatment is to begin six weeks following patient ESD/EMR surgery.
  Patients may delay dosing under the following certain circumstances:
  1. Dosing may be delayed per Toxicity Management Guidelines (Appendix IV), due to either an immune or a non-immune-related AE.
  2. Dosing intervals of subsequent cycles may be shortened as clinically feasible in order to gradually align treatment cycles with the schedule of tumor efficacy (RECIST) and PRO assessments. Subsequent time between 2 consecutive doses cannot be less than 22 days, based on the half-lives of durvalumab (see current Investigator Brochure for durvalumab).
  3. Standard of Care Arm (CROSS):
  4. Patients may delay and subsequently resume dosing per local standard clinical practice.
  If dosing must be delayed for reasons other than treatment-related toxicity, dosing will occur as soon as feasible.
  Arms: Adjuvant Immunoradiotherapy (ARM1) and Adjuvant Immunotherapy (ARM1B)
Drug: Adjuvant chemoradiotherapy — Durvalumab treatment is to begin six weeks following patient ESD/EMR surgery.
  Patients may delay dosing under the following certain circumstances:
  1. Dosing may be delayed per Toxicity Management Guidelines (Appendix IV), due to either an immune or a non-immune-related AE.
  2. Dosing intervals of subsequent cycles may be shortened as clinically feasible in order to gradually align treatment cycles with the schedule of tumor efficacy (RECIST) and PRO assessments. Subsequent time between 2 consecutive doses cannot be less than 22 days, based on the half-lives of durvalumab (see current Investigator Brochure for durvalumab).
  3. Standard of Care Arm (CROSS):
  4. Patients may delay and subsequently resume dosing per local standard clinical practice.
  If dosing must be delayed for reasons other than treatment-related toxicity, dosing will occur as soon as feasible.
  Arms: Adjuvant chemoradiotherapy

SUMMARY:
The goal of this study is to assess the safety of delivering concurrent adjuvant chemoradiation or immuno-radiation therapy after EMR/ESD in pT1b/T2N0 esophageal cancer patients. The main objectives of the study are:

1. Assess the feasibility of enrolling 10 patients.
2. Assess the safety of delivering concurrent adjuvant chemoradiation or immunoradiation therapy after EMR/ESD in pT1b/T2 esophageal cancer patients

DETAILED DESCRIPTION:
This is a single center trial to assess feasibility and safety of conducting a multicenter Phase I non-randomized trial of adjuvant Durvalumab therapy in the treatment of pT1b/T2N0 esophageal cancer. The investigatory treatment, ARM1, will be endoscopic resection followed by adjuvant immunoradiation therapy. Patients that are recruited but are unable to receive immunotherapy will be recruited to ARM2 the current standard of care in chemoradiation therapy The study will include patients diagnosed with pT1b/T2 esophageal cancer after endoscopic resection that are ineligible for an esophagectomy or for those who decline an esophagectomy as treatment.

The current standard of care for treatment of pT1b/T2 esophageal cancer is esophagectomy with postoperative adjuvant chemotherapy. Depending on the detection of nodal metastasis during intraoperative nodal sampling, patients that are truly N0 can avoid postoperative adjuvant chemotherapy. Patients that are ineligible for esophagectomy or decline an esophagectomy as treatment are directed to concurrent chemoradiation (Table ESOPH-F, Adjani et al. 2019). Combined modality chemoradiation therapy, paclitaxel and carboplatin concurrent with radiation therapy (50 to 50.4 Gy) is classified as Category One treatment regime according to the most current CROSS protocol (van Hagen et al. 2012). Chemoradiation is the recommended first-line of preoperative treatment for patients that can tolerate an esophagectomy (ESOPH-F). It is also recommended as the first-line of concurrent treatment for localized esophageal cancers that are ineligible for esophagectomy (ESOPH-17). In the current standard of treatment, patients that are ineligible for esophagectomy or decline an esophagectomy and cannot tolerate chemoradiation are directed to radiation therapy as a palliative treatment. The goal of the current study is to provide a curative multi-modal option to patients that are ineligible for esophagectomy and to provide an alternative systemic therapy for patients that are not candidates for the current standard in multimodal treatments such as chemoradiation therapy. Patients may be considered ineligible for esophagectomy due to 1) inoperability of the tumour due to location, 2) the patient is considered high risk for serious intra-operative or post-operative complications and 3) patients may decline an esophagectomy as a line of treatment. Esophagectomy is a complicated surgical procedure associated with serious intraoperative and postoperative complications. Loss of organ function can result in life-long risk of complications. Endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) is currently routinely performed as a diagnostic and sampling procedure. The current study will determine the therapeutic and quality of life benefits of ESD/EMR in combination with systemic monotherapy and radiation therapies in a patient population that is ineligible for esophagectomy. The current study will assess feasibility of patient recruitment over an 18 month period and safety profile of Durvalumab as an adjuvant treatment within this patient population.

In patients with early-stage esophageal cancer with clinical T1 or T2N0 stage, clinical staging alone is unreliable. EMR/ESD is done both as a diagnostic and potentially curative procedure. EMR/ESD will identify if a patient truly has pT1 or pT2 disease. In patients with fully resected pT1a or low risk pT1b cancer (i.e., resected via EMR/ESD), adjuvant treatment is not indicated and would be considered to have greater risks than benefits. Thus, pursuing a neo-adjuvant therapy approach (i.e. giving immunoradiation therapy before EMR/ESD) should be avoided for the following reasons: 1) it would obscure the true pathologic stage of the cancer 2) it would make the EMR/ESD more complicated due to submucosal fibrosis and would thus increase the risks of complications 3) it would put people through treatments they would never have needed and would only confer risks rather than benefits (i.e. patients with fully resected pT1a or low-risk pT1b cancer).

ELIGIBILITY:
Inclusion Criteria:

* AGE >18
* Able to provide informed consent.
* Pathological stage T1B or T2 esophageal or non-metastatic gastro-esophageal adenocarcinoma, squamous cell cancer or mixed histology.
* Ineligible for or declining esophagectomy.
* Completed endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD).
* Body weight >30kg
* Adequate normal organ and marrow function as defined below:

  1. Haemoglobin ≥9.0 g/dL
  2. Absolute neutrophil count (ANC) ≥1.0 × 109 /L
  3. Platelet count ≥75 × 109/L
  4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
  5. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
  6. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks

Exclusion Criteria:

* • Participation in another clinical study with an investigational product during the last 4 weeks.

  * Concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
  * Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) ≤15 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca and the investigator.
  * Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia and vitiligo.

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
  * Any concurrent chemotherapy, investigative product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
  * Radiotherapy treatment to more than 30% of the bone marrow within 4 weeks of the first dose of study drug.
  * Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of durvalumab. Note: Local surgery of isolated lesions for palliative intent is acceptable.
  * History of allogenic organ transplantation.
  * Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia.
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
    3. Any chronic skin condition that does not require systemic therapy.
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
    5. Patients with celiac disease controlled by diet alone.
  * Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
  * History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of durvalumab and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
  * History of leptomeningeal carcinomatosis
  * Patients with brain or any other brain metastases
  * History of active primary immunodeficiency
  * Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  * Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
  * Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab.
  * Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
  * Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
  * Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
  * Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
  * Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of enrolling 10 patients | 1.5 years
  Assess the feasibility of enrolling 10 patients (i.e. Raw count of number of patients enrolled in 1.5 years)
Safety (proportion of patients developing Grade 3 or above adverse events) | 1.5 years
  Assess the safety of delivering concurrent adjuvant chemoradiation or immunoradiation therapy after EMR/ESD in pT1b/T2 esophageal cancer patients. This will be done using CTCAE. This will be descriptive and be based on proportion of patients developing Grade 3 or above adverse events.

SECONDARY OUTCOMES:
Health-related quality of life (change in FACT-E score between pretreatment/baseline score to the score at the 2-year mark post-resection) | 2 years
  Determine health-related quality of life, based on longitudinal assessment of validated FACT-E scale (Functional Assessment of Cancer Therapy - Esophageal). This will be descriptive and be based on the change from pretreatment/baseline score to the score at the 2-year mark post-resection. FACT-E has 44 questions scored on a 5-point Likert scale, with lower scoring indicating less effects on quality of life.
Progression-free survival | 2 years
  Determine progression-free survival at 2 years, using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Biniam Kidane, Principal Investigator — University of Manitoba
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No